CLINICAL TRIAL: NCT00942266
Title: A Randomized Phase II Study of Two Dose-Levels of Vorinostat in Combination With 5-FU and Leucovorin in Patients With Refractory Metastatic Colorectal Cancer
Brief Title: Vorinostat, Fluorouracil, and Leucovorin Calcium in Treating Patients With Metastatic Colorectal Cancer That Has Not Responded to Previous Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 142808; NCI-2009-01523
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-05

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive low-dose oral vorinostat once daily on days 1-3, leucovorin calcium IV over 2 hours on day 2, and fluorouracil IV over 46 hours on days 2 and 3. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: vorinostat; Other: pharmacological study
- Arm II (Experimental): Patients receive high-dose oral vorinostat once daily on days 1-3 and leucovorin calcium and fluorouracil as in arm I. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: vorinostat; Other: pharmacological study

INTERVENTIONS:
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU; Adrucil; Efudex; FU
Drug: leucovorin calcium — Given IV
  Other Names: calcium folinate; CF; CFR; citrovorum factor; LV; Wellcovorin
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: pharmacological study — Correlative study
  Other Names: pharmacological studies

SUMMARY:
RATIONALE: Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as fluorouracil and leucovorin calcium, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known which dose of vorinostat is more effective when given together with combination chemotherapy in treating patients with metastatic colorectal cancer. PURPOSE: This randomized phase II trial is studying the best dose of vorinostat to see how well it works when given together with fluorouracil and leucovorin calcium in treating patients with metastatic colorectal cancer that has not responded to previous treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. Describe the 2-months progression free rate on vorinostat 800mg/day x 3 in combination with 5-FU/L V every 2 weeks. (Arm I) II. Describe the 2-months progression free rate on vorinostat 1400mg/day x 3 in combination with 5-FU/L V every 2 weeks. (Arm II) SECONDARY OBJECTIVES: I. Describe the response rate on Arm 1 and Arm 2 of the study. II. Estimate the median progression free survival on both arms of the study. III. Describe the overall survival on Arm 1 and Arm 2 of the study. IV. Describe the toxicities on Arm 1 and Arm 2 of the study. V. Describe vorinostat pharmacokinetics on Arm 1 and Arm 2 of the study. VI. Describe 5-FU steady state pharmacokinetics on Arm 1 and Arm 2 of the study. OUTLINE: Patients are randomized to 1 of 2 treatment arms. ARM I: Patients receive low-dose oral vorinostat once daily on days 1-3, leucovorin calcium IV over 2 hours on day 2, and fluorouracil IV over 46 hours on days 2 and 3. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. ARM II: Patients receive high-dose oral vorinostat once daily on days 1-3 and leucovorin calcium and fluorouracil as in arm I. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity. After completion of study therapy, patients are followed up for 30 days and then every 3 months.

ELIGIBILITY:
Inclusion

* Patients must have histologically or cytologically confirmed colorectal adenocarcinoma that is metastatic and which has failed standard treatment or for which no standard treatment is available
* Patients should have fluoropyrimidine-refractory disease; radiographic evidence of progression within 4 weeks from the last dose of a fluoropyrimidine-based regimen (at least 6 weeks of fluoropyrimidine-based treatment)
* Patients should have received and progressed on (or proved to be intolerant to) oxaliplatin and irinotecan; progression within 6 months from oxaliplatin-based therapy or irinotecan-based therapy is acceptable for eligibility
* Patients with KRAS wild-type or unknown KRAS status tumors should have progressed on or within 6 months from last cetuximab or panitumumab-based therapy; no prior cetuximab therapy is required for KRAS mutant tumors
* ECOG performance status =< 2
* Life expectancy >= 12 weeks
* Ability to understand and the willingness to sign a written informed consent document
* Ability to swallow pills
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< institutional upper limit of normal
* AST(SGOT)/ALT(SGPT) =< 3 x institutional upper limit of normal in the absence of metastatic disease to the liver and =< 5 x institutional upper limit of normal in the setting of metastatic disease to the liver
* Creatinine =< 1.5 x institutional upper limit of normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Males undergoing study treatment should also agree to adequate measures of contraception (partner contraception and use of condoms or abstinence, or vasectomy)

Exclusion

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from significant adverse events due to agents administered more than 3 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat or other agents used in study
* Greater than Grade 2 neuropathy as defined by CTCAE version 3.0
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Baseline EKG with QTc prolongation that is grade 2 or higher by CTCAE version 3.0
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with vorinostat
* Patients should not have taken valproic acid or other histone deacetylase inhibitors, for at least 4 weeks prior to enrollment
* Patients with known HIV infection or known active viral hepatitis
* Prior treatment with vorinostat
* Other non-study medications known to increase the QTc interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-07; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen Wee MA, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Low-dose Vorinostat: Patients receive low-dose oral vorinostat once daily on days 1-3, leucovorin calcium IV over 2 hours on day 2, and fluorouracil IV over 46 hours on days 2 and 3. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
  fluorouracil: Given IV
  leucovorin calcium: Given IV
  vorinostat: Given orally
  pharmacological study: Correlative study
- Arm II: High-dose Vorinostat: Patients receive high-dose oral vorinostat once daily on days 1-3 and leucovorin calcium and fluorouracil as in arm I. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
  fluorouracil: Given IV
  leucovorin calcium: Given IV
  vorinostat: Given orally
  pharmacological study: Correlative study
Period: Overall Study
Arm/Group | Arm I: Low-dose Vorinostat | Arm II: High-dose Vorinostat
Started | 43 | 15
Completed | 0 | 0
Not Completed | 43 | 15
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 2 | 1
Not completed — Disease Progression | 38 | 11
Not completed — Failure to thrive and pt withdrawal | 0 | 1
Not completed — Intercurrent illness | 0 | 1
Not completed — Physician Decision | 2 | 0
Not completed — medical deterioration (pneumonia) | 0 | 1

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients; per protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Low-dose Vorinostat | Arm II: High-dose Vorinostat | Total
Number analyzed (Participants) | 43 | 15 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (10.3) | 61.1 (10.5) | 60.6 (10.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 9 | 38
  >=65 years | 14 | 6 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 9 | 31
  Male | 21 | 6 | 27

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (Stable Disease or Objective Response)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI:
  Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: At 2 months
Population: All treated and eligible patients; per protocol
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I: Low-dose Vorinostat | Arm II: High-dose Vorinostat
Number analyzed (Participants) | 43 | 15
percentage of participants | 53 [38 to 68] | 53 [28 to 78]

2. Secondary Outcome: Median Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Every 8 weeks, up to 100 weeks.
Population: All treated and eligible patients; per protocol
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: Low-dose Vorinostat | Arm II: High-dose Vorinostat
Number analyzed (Participants) | 43 | 15
months | 2.4 [1.8 to 3.6] | 2.9 [1.6 to 5.6]

3. Secondary Outcome: Response Rate
Description: as for outcome 1
Time Frame: Every 8 weeks; up to 100 weeks.
Population: All treated and eligible patients; per protocol
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I: Low-dose Vorinostat | Arm II: High-dose Vorinostat
Number analyzed (Participants) | 43 | 15
percentage of participants | 2.3 [0 to 6.8] | 100 [100 to 100]

4. Secondary Outcome: Toxicity
Description: Number of participants with an adverse event.
  Please refer to the adverse event reporting for more detail.
Time Frame: Daily
Population: All treated and eligible patients; per protocol
Measure: Number; unit: participants
Arm/Group | Arm I: Low-dose Vorinostat | Arm II: High-dose Vorinostat
Number analyzed (Participants) | 43 | 15
participants | 42 | 15

5. Secondary Outcome: Overall Survival
Time Frame: Every 12 weeks
Population: All treated and eligible patients; per protocol
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I: Low-dose Vorinostat | Arm II: High-dose Vorinostat
Number analyzed (Participants) | 43 | 15
months | 6.5 [4.8 to 7.8] | 6.7 [3.0 to 21.9]

6. Secondary Outcome: Vorinostat Pharmacokinetics
Description: Blood samples (5 ml of blood each) will be collected in red-top vacutainers (no anticoagulant) at 0 (pre- vorinostat), 0.5, 1, 2, 3, 4, 6, and 8 hours after the vorinostat dose on the first day of 5-FU infusion on cycle 1 (day 2 of cycle 1). Mean area under the curve is presented with 95% CI.
Time Frame: day 2 (cycle 1)
Population: Vorinostat PKs were be performed on day 2 of vorinostat in the first 10 patients of each arm treated at RPCI
Measure: Mean (95% Confidence Interval); unit: hr∙μM
Arm/Group | Arm I: Low-dose Vorinostat | Arm II: High-dose Vorinostat
Number analyzed (Participants) | 10 | 10
hr∙μM | 12.6 [4.9 to 38.4] | 14.7 [4.5 to 42.7]

7. Secondary Outcome: Fluorouracil Steady-state Pharmacokinetics
Description: Blood samples will be collected for determination of plasma 5-FU steady state concentration at 6 hours after start of 5-FU continuous infusion. The mean per treatment arm are presented.
Time Frame: Day 1
Population: All treated and eligible patients
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Arm I: Low-dose Vorinostat | Arm II: High-dose Vorinostat
Number analyzed (Participants) | 12 | 15
ng/ml | 389.4 [328.9 to 449.9] | 423.5 [339.0 to 508.0]

ADVERSE EVENTS:
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 12/43 | 6/15
Other Adverse Events (participants affected / at risk) | 42/43 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=43) | Arm II (N=15)
Tachycardia (Cardiac disorders) | 1 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (4) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (4) | 1 (4)
Nausea (Gastrointestinal disorders) | 2 (15) | 1 (4)
Vomiting (Gastrointestinal disorders) | 2 (12) | 1 (8)
Cholangitis (Hepatobiliary disorders) | 1 (4) | 0 (0)
Infection (Infections and infestations) | 1 (8) | 1 (4)
Pneumonia (Infections and infestations) | 1 (4) | 1 (4)
Troponin I increased (Investigations) | 1 (4) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Convulsion (Nervous system disorders) | 1 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (8) | 0 (0)
Hypotension (Vascular disorders) | 1 (4) | 1 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=43) | Arm II (N=15)
Anaemia (Blood and lymphatic system disorders) | 10 (51) | 2 (7)
Leukopenia (Blood and lymphatic system disorders) | 5 (24) | 1 (4)
Lymphopenia (Blood and lymphatic system disorders) | 11 (55) | 7 (74)
Neutropenia (Blood and lymphatic system disorders) | 2 (8) | 3 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (4) | 1 (4)
Tachycardia (Cardiac disorders) | 1 (8) | 0 (0)
Cataract (Eye disorders) | 1 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (4) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 3 (12) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (3) | 1 (4)
Dental caries (Gastrointestinal disorders) | 1 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (24) | 1 (4)
Dyspepsia (Gastrointestinal disorders) | 5 (20) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (8)
Nausea (Gastrointestinal disorders) | 12 (63) | 9 (40)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (4)
Stomatitis (Gastrointestinal disorders) | 2 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (24) | 2 (8)
Fatigue (General disorders) | 11 (72) | 5 (36)
Mucosal inflammation (General disorders) | 4 (16) | 3 (24)
Oedema peripheral (General disorders) | 1 (4) | 0 (0)
Pain (General disorders) | 3 (12) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (8) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (8) | 0 (0)
Cystitis (Infections and infestations) | 1 (3) | 0 (0)
Herpes virus infection (Infections and infestations) | 1 (8) | 0 (0)
Infection (Infections and infestations) | 1 (4) | 0 (0)
Localised infection (Infections and infestations) | 1 (4) | 0 (0)
Sinusitis (Infections and infestations) | 1 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (4) | 0 (0)
Vaginitis bacterial (Infections and infestations) | 0 (0) | 1 (4)
Fracture (Injury, poisoning and procedural complications) | 1 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (8) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (20) | 3 (12)
Blood albumin decreased (Investigations) | 1 (4) | 0 (0)
Blood alkaline phosphatase (Investigations) | 1 (4) | 1 (4)
Blood alkaline phosphatase increased (Investigations) | 2 (8) | 3 (12)
Blood creatinine increased (Investigations) | 1 (4) | 1 (7)
Blood thyroid stimulating hormone increased (Investigations) | 1 (3) | 0 (0)
Electrocardiogram QT corrected interval (Investigations) | 0 (0) | 1 (4)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 4 (17)
Haemoglobin decreased (Investigations) | 1 (8) | 4 (32)
International normalised ratio increased (Investigations) | 0 (0) | 1 (4)
Lipase increased (Investigations) | 1 (4) | 0 (0)
Troponin I increased (Investigations) | 1 (4) | 0 (0)
Urine colour abnormal (Investigations) | 1 (4) | 0 (0)
Weight decreased (Investigations) | 2 (8) | 1 (4)
Anorexia (Metabolism and nutrition disorders) | 10 (48) | 5 (20)
Dehydration (Metabolism and nutrition disorders) | 3 (12) | 1 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (28) | 4 (28)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (23) | 2 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (24) | 2 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (12) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (16) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Convulsion (Nervous system disorders) | 1 (4) | 0 (0)
Dizziness (Nervous system disorders) | 1 (4) | 1 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (12)
Headache (Nervous system disorders) | 0 (0) | 1 (4)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (4)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (4)
Anxiety (Psychiatric disorders) | 1 (4) | 0 (0)
Depression (Psychiatric disorders) | 1 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (8) | 1 (4)
Enuresis (Renal and urinary disorders) | 1 (4) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (4)
Pollakiuria (Renal and urinary disorders) | 1 (4) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (11) | 1 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (8) | 1 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (8) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (24) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (16) | 0 (0)
Hypertension (Vascular disorders) | 1 (4) | 0 (0)
Phlebitis superficial (Vascular disorders) | 1 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes